CLINICAL TRIAL: NCT01984086
Title: An Open-label, Randomised, Cross-over, Two Cohort, Single Dose Study in Healthy Volunteers to Evaluate the Unit Dose Dry Powder Inhaler (UD-DPI) for the Delivery of Salbutamol and to Compare the Pharmacokinetic Profile With the MDI and Diskus Presentations.
Brief Title: Study to Evaluate the Pharmacokinetic Profile of Salbutamol Delivered by Unit Dose Dry Powder Inhaler (UD-DPI) Compared to the Diskus and Metered Dose Inhaler (MDI) in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200921
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: COPD; Asthma; Respiratory
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Subjects will receive following six treatments each in six period, with a 3-days minimum wash-out period, between each treatment period: 1) Single dose (SD) salbutamol (200mcg per blister from 1.6% blend) delivered via the UD-DPI by inhalation of 3 Blisters (BTR) giving a total dose of 600mcg; 2) SD salbutamol sulphate (200mcg per BTR from a 1.0% blend) delivered via the UD-DPI by inhalation of 3 BTR giving a total dose of 600mcg; 3) SD salbutamol (150mcg per BTR from a 1.6% blend) delivered via the UD-DPI by inhalation of 3 BTR giving a total dose of 450mcg; 4) SD salbutamol (250mcg per BTR from a 1.6% blend) delivered via the UD-DPI by inhalation of 3 BTR giving a total dose of 750mcg; 5) SD of salbutamol (200mcg per BTR) delivered via the Diskus by inhalation of 3 BTR giving a total dose of 600mcg; 6) SD salbutamol (100mcg per actuation) delivered via the MDI giving a total dose of 600mcg
  Interventions: Drug: Salbutamol Sulphate 150mcg UD-DPI Blister(1.6% blend); Drug: Salbutamol Sulphate 200mcg UD-DPI Blister(1.6% blend); Drug: Salbutamol Sulphate 250mcg UD-DPI Blister(1.6% blend); Drug: Salbutamol Sulphate 200mcg UD-DPI Blister(1% blend); Drug: Salbutamol Diskus 200mcg Blister; Drug: Salbutamol MDI 100mcg
- Part B (Experimental): Prior to the start of Part B, a decision will be made regarding the UD-DPI products to be used in Part B. Subjects will receive following 6 treatments each in 6 period, with a 3-days minimum wash-out period, between each treatment period: 1) SD salbutamol (selected from Part A) delivered via the UD-DPI without activated charcoal (AC) by inhalation of 3 BTR (total dose dependant on UD-DPI formulation chosen); 2) SD salbutamol (selected from Part A) delivered via the UD-DPI with AC by inhalation of 3 BTR (total dose dependant on UD-DPI formulation chosen); 3) SD salbutamol by inhalation of 3 BTR (200mcg per BTR) delivered via the Diskus without AC (total dose 600mcg); 4) SD salbutamol by inhalation of 3 BTR (200mcg per BTR) delivered via the Diskus with AC (total dose 600mcg); 5) SD salbutamol 6 inhalations (100mcg) delivered via the MDI without AC (total dose 600mcg); 6) SD salbutamol 6 inhalations (100mcg) delivered via the MDI with AC (total dose 600mcg)
  Interventions: Drug: Salbutamol Sulphate UD-DPI Blister (selected from Part A); Drug: Salbutamol Sulphate 250mcg UD-DPI Blister (selected from Part A); Drug: Salbutamol Diskus 200mcg Blister without activated charcoal; Drug: Salbutamol Diskus 200mcg Blister with activated charcoal; Drug: Salbutamol MDI 100mcg without activated charcoal; Drug: Salbutamol MDI 100mcg with activated charcoal

INTERVENTIONS:
Drug: Salbutamol Sulphate 150mcg UD-DPI Blister(1.6% blend) — Salbutamol Sulphate 150mcg UD-DPI will be supplied as blister containing a small quantity of powder comprising of a blend of salbutamol sulphate (micronized) and excipients
  Arms: Part A
Drug: Salbutamol Sulphate 200mcg UD-DPI Blister(1.6% blend) — Salbutamol Sulphate 200mcg UD-DPI will be supplied as blister containing a small quantity of powder comprising of a blend of salbutamol sulphate (micronized) and excipients
  Arms: Part A
Drug: Salbutamol Sulphate 250mcg UD-DPI Blister(1.6% blend) — Salbutamol Sulphate 250mcg UD-DPI will be supplied as blister containing a small quantity of powder comprising of a blend of salbutamol sulphate (micronized) and excipients
  Arms: Part A
Drug: Salbutamol Sulphate 200mcg UD-DPI Blister(1% blend) — Salbutamol Sulphate 200mcg UD-DPI will be supplied as blister containing a small quantity of powder comprising of a blend of salbutamol sulphate (micronized) and excipients
  Arms: Part A
Drug: Salbutamol Diskus 200mcg Blister — Salbutamol Diskus 200mcg will be supplied as blister strip contained within the Diskus device. Each blister contains a small quantity of powder comprising of a blend of salbutamol sulphate (micronized) and excipients
  Arms: Part A
Drug: Salbutamol MDI 100mcg — Salbutamol MDI 100mcg will be supplied as formulation of salbutamol sulphate (micronized) in propellant contained within the pressurised MDI device
  Arms: Part A
Drug: Salbutamol Sulphate UD-DPI Blister (selected from Part A) — Formulation will be determined depending on the outcome of Part A.
  Arms: Part B
Drug: Salbutamol Sulphate 250mcg UD-DPI Blister (selected from Part A) — Formulation will be determined depending on the outcome of Part A.
  Arms: Part B
Drug: Salbutamol Diskus 200mcg Blister without activated charcoal — Formulation will be determined depending on the outcome of Part A.
  Arms: Part B
Drug: Salbutamol Diskus 200mcg Blister with activated charcoal — Formulation will be determined depending on the outcome of Part A.
  Arms: Part B
Drug: Salbutamol MDI 100mcg without activated charcoal — Formulation will be determined depending on the outcome of Part A.
  Arms: Part B
Drug: Salbutamol MDI 100mcg with activated charcoal — Formulation will be determined depending on the outcome of Part A.
  Arms: Part B

SUMMARY:
This is an open-label, two part, six period- cross over, randomised, single dose, single centre study in healthy subjects. This is the first clinical study for the UD-DPI. This study is divided into two parts. Part A will ascertain whether the pharmacokinetic (PK) of salbutamol delivered via the UD-DPI is comparable to the salbutamol delivered via the Diskus or MDI. For this reason four treatment doses consisting of three dose strength and two percentage blends will be assessed in Part A delivered via UD-DPI. Part A will also provide preliminary PK variability estimates to allow for better sample size/precision calculations for Part B. Part B will explore whether the UD-DPI has a pharmacokinetic exposure profile that is comparable to either Diskus or MDI in the presence of the charcoal block.

ELIGIBILITY:
Inclusion Criteria

* Male/females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight >=50 kg and body mass index within the range 19.0 - 34.0 kilogram per square meter (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli-international units per milliliter (MlU/mL) and estradiol < 40 picograms per milliliter (pg/mL) (<147 picomole per liter) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in listed in protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential with negative pregnancy test as determined by serum human chorionic gonadotropin (hCG) test at screening or urine hCG prior to dosing AND; Agrees to use one of the contraception methods listed in protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until follow-up; OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Alanine transaminase, alkaline phosphatase and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate ECGs obtained over a brief recording period: QTcF <450 milliseconds.
* Current non-smokers who have not used any tobacco- containing products within 3 months of screening and with a total pack year history of <=10 pack years [number of pack years = (number of cigarettes per day / 20) x number of years smoked].
* Able to use all medical device products included in the study adequately after training

Part B

* Able to tolerate the charcoal block at screening

Exclusion Criteria

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of sensitivity to any of the study medications, or components thereof (including milk protein allergy) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study breath carbon monoxide test or urine drug or breath alcohol screen.
* A positive test for HIV antibody.
* Screening PR interval outside the range 120 to 240msec; or an ECG that is not suitable for QT measurements (eg poorly defined termination of T-wave)
* Pregnant or lactating females or females actively trying to conceive.
* Where participation in the study would result in donation of blood or blood products in excess of 500 millilitres within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* An unwillingness to abstain from strenuous exercise starting 72 hours prior to each dosing day
* An unwillingness to abstain from caffeine- and xantheine- containing products for 24 hours prior to dosing.
* Subject is mentally or legally incapacitated

Part B

* Previous participation in Part A of this study (200921)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2014-05-26 (Actual); Study Completion 2014-05-26 (Actual)

PRIMARY OUTCOMES:
Part A: Pharmacokinetics parameters of single doses of salbutamol in healthy subjects delivered via the UD-DPI device, using a range of doses and blends, and to compare to MDI and Diskus | Day 1 of each treatment period (Pre dose and 0 hr, 2 minute [min], 5 min, 10 min, 20 min, 30 min, 45 min, 1hr, 1.5 hr, 2hr, 4 hr, 6 hr, 8 hr, 10 hr and 12 hr post dose)
  PK parameters include: area under the concentration-time curve from time zero (pre-dose) to 12 hours (hr) (AUC [0-12hr]) and/ or area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-infinity]) and/ or area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC [0-t]) and maximum observed concentration (Cmax).
Part B: Pharmacokinetics parameters of salbutamol in healthy subjects delivered via UD-DPI versus Diskus and/or MDI with charcoal blockade. | Day 1 of each treatment period (Pre dose and 0 hr, 2 minute [min], 5 min, 10 min, 20 min, 30 min, 45 min, 1hr, 1.5 hr, 2hr, 4 hr, 6 hr, 8 hr, 10 hr and 12 hr post dose)
  PK parameters include: AUC(0- infinity) or AUC(0-t) and Cmax

SECONDARY OUTCOMES:
Part A: Pharmacokinetic parameters following single doses of salbutamol and different blends of salbutamol in healthy subjects delivered via UD-DPI | Day 1 of each treatment period (Pre dose and 0 hr, 2 minute [min], 5 min, 10 min, 20 min, 30 min, 45 min, 1hr, 1.5 hr, 2hr, 4 hr, 6 hr, 8 hr, 10 hr and 12 hr post dose)
  PK parameters include: area under the concentration-time curve from time zero (pre-dose) to 30 min (AUC [0-30 min]) and time to maximum observed concentration (tmax).
Part B: Pharmacokinetic parameters following single doses of salbutamol in healthy subjects delivered via UD-DPI , MDI and Diskus with/ and without charcoal | Day 1 of each treatment period (Pre dose and 0 hr, 2 minute [min], 5 min, 10 min, 20 min, 30 min, 45 min, 1hr, 1.5 hr, 2hr, 4 hr, 6 hr, 8 hr, 10 hr and 12 hr post dose)
  PK parameters include: AUC [0 30 min] and tmax
Part A and B: Number of subjects with adverse events (AEs) | Up to 14 days after the last dose of study treatment.
Part A and B: Safety and tolerability of salbutamol, as assessed vital signs | Day 1 of each treatment period
  Vital sign measurements to be measurement include systolic and diastolic blood pressure and pulse rate
Part A and B: Safety and tolerability of salbutamol, as assessed by 12-lead electrocardiogram (ECG) parameters | Day 1 of each treatment period
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT interval using Fredericia's formula (QTcF) intervals.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200921 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200921?search=study&search_terms=200921#rs
- Available data/document: Clinical Study Report: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200921 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register